CLINICAL TRIAL: NCT06547970
Title: The Impact of Pharmacist Led Education Program on Glycemic Control, Quality of Life and Medication Adherence Among Patients With Type 1 Diabetes Mellitus
Brief Title: Pharmacist Led Educational Intervention on QOL, Medication Adherence & Satisfaction on Patients With Type 1 DM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Marwah Salman Abdulrahman, clinical pharmacist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DM type 1
Record Dates: First submitted 2024-07-24; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (no education) (Placebo Comparator): a group of DM patients we will record their HbA1C , FBG & their QOL by filling the questionnaire (will be filled by the researcher herself then after 3 months we are going to record the same variables
  Interventions: Other: Educational intervension
- Patient education (Active Comparator): a group of DM patients we will record their HbA1C , FBG & their QOL, medication adherence , insulin taking technique form ( the questionnaire & form will be filled by the researcher herself) then an educational session will last about 30 min. will be given to each patient face to face at the last the recearcherr and the patients will share their phone numbers for following up then after 3 months all the variables will be recorded again
  Interventions: Other: Educational intervension

INTERVENTIONS:
Other: Educational intervension — an educational intervention about the disease, symptoms & how to deal with these symptoms, foot care, life style like sport and nutritional advices
  Other Names: follow up

SUMMARY:
There was no previous study in Iraq to evaluate the efficacy of pharmacist-led educational intervention on patient glycemic control, quality of life and medication adherence among type 1 diabetic patients in Iraq.

Improving diabetes patients' information's about their disease control, the role of insulin and the right technique to administer it, how to deal with hyper- and hypoglycemia, about their diet and exercise.

It is important to conduct a study to evaluate the pharmacist's role in education and improving patients' quality of life.

DETAILED DESCRIPTION:
Aim of the Study:

The aim of the current study is to evaluate the impact of pharmacist-led educational intervention on glycemic control, quality of life and medication adherence among type 1 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* - Patients age ≥ 16 years old who can speak and read the Arabic language.
* Had been diagnosed with T1DM for at least 6 months ago.
* Had uncontrolled hyperglycemia (glycosylated hemoglobin HbA1C ≥7% and/or fasting blood glucose >130 mg/dl)
* Patients on the same regimen the last 3 months.
* patients (or parents) acceptance to participate in the study.

Exclusion Criteria:

* 1-Patient who have hearing, speech or cognitive deficits that would impair understanding of the questions and receiving the education.

  2- Patients with comorbid conditions that may interfere with the study such as asthma, thyroid disorders, adrenal gland disorders, celiac disease, or significant renal impairment.

  3-Patients who are taking corticosteroids. 4- Patients who required changing their insulin regimen, increasing the dose >20% of the previous dose. (21) 5- Patients with conditions that affect red blood cell turnover (hemolytic and other anemias, G-6-PD deficiency, recent blood transfusion, use of drugs that stimulate erythropoiesis, end stage kidney disease and pregnancy.

  6-Patients unwilling to participate.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin A1c (%) (HbA1c) | Baseline (beginning of the intervention) and the end of 3 months follow-up.
  Measurement of Glycated hemoglobin A1c (%) (HbA1c) at beginning of the intervention and the end of 3 months follow-up.
The Quality of Life Scale (QoL) | Baseline (beginning of the intervention) and the end of 3 months follow-up.
  The score consists of four major domains including general health, social, psychological, and satisfaction issues. Ten items were selected to formulate the quality-of-life scale for Iraqi DM patients (QOLSID). The first four questions with question ten are used to directly assess satisfaction, question five is used to assess social issue while questions six and seven were used to assess emotion and stress finally question eight and nine are directly used to assess health issue. The score of each question range from 0 (poor) to 5 (optimum). Items 1,2,6 and 7 with reverse scoring. Total score = direct summation of all items scores. Total scores ≥ 32.5 points refer to good quality of life.

SECONDARY OUTCOMES:
Anti-Diabetic Medication Adherence Scale (IADMAS) | Baseline (beginning of the intervention) and the end of 3 months follow-up.
  The scale consists of eight items; three items are used to directly assess medication-taking behavior by giving five responses: (1) always (daily), (2) often, (3) sometimes, (4) rarely and (5) never. The remaining five items are used to measure the determinant of non-adherence by giving a dichotomous response of "Yes" or "No". The first item aims to identify the extent of unintentional missing of medication doses; all other questions were directed to identify the extent of intentional medication non-adherence. Two items (1 and 3) were used to identify the extent of non-adherence to the time of medication taking. Four items (2, 6, 7 and 8) were formulated to identify the extent of intentional non-adherence with the prescribed medication dose. Only one item (5) aims to identify the extent of intentional non-adherence through discontinuation of taking DM medication. Scoring of all items ranged from 0 to 1, 0 for non-adherent answer and 1 for total adherence.
Insulin self-administration assessment checking list | Baseline (beginning of the intervention) and the end of 3 months follow-up.
  The assessment form was developed based on the latest expert recommendations for best practice in insulin injection technique. to assess pharmacists' counseling and educational role about the use of insulin. Areas of assessment include Preparations for injecting insulin contain six questions, Insulin injecting technique contain nine questions, Storage and stability of insulin contain 2 questions. the answers would be yes and no

CONTACTS AND LOCATIONS:
Overall Officials: Ali Lateef Jasim, PhD, Study Director — Baghdad University
Locations (1):
- Al-kindy Specialized center for endocrine diseases and diabetes, Baghdad, Iraq